CLINICAL TRIAL: NCT06813287
Title: Brain Monitoring, tDCS and Robotic Training in SCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kathleen Friel (Other)
Responsible Party: Sponsor-Investigator, Kathleen Friel, Lab Director, Clinical Laboratory for Early Brain Injury Recovery, Burke Medical Research Institute
Organization: Burke Medical Research Institute (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BRC442
Record Dates: First submitted 2018-05-17; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS & EEG (Experimental): 20 minutes of real anodal tDCS of cortical neurophysiology and EEG responses in chronic spinal cord injury patients.
  Interventions: Diagnostic Test: Electroencephalography (EEG)
- Sham tDCS (Sham Comparator): 2 weeks (5x per week) of upper limb robotic training in conjunction with sham tDCS.
  Interventions: Device: Upper extremity robot
- Active tDCS (Experimental): 2 weeks (5x per week) of upper limb robotic training in conjunction with active tDCS.
  Interventions: Device: Upper extremity robot

INTERVENTIONS:
Diagnostic Test: Electroencephalography (EEG) — Recording of electrical activity in the brain
  Arms: tDCS & EEG
Device: Upper extremity robot — Used for training and objective assessment (kinematics)
  Arms: Active tDCS; Sham tDCS

SUMMARY:
To explore the neurophysiological and electroencephalography (EEG) changes that one single session of tDCS and robotics has in the SCI population (Study 1); and to investigate upper limb motor recovery in chronic tetraplegia SCI patients, comparing two rehabilitation strategies: real or sham tDCS combined with upper-limb robotic therapy (Study 2), as well as to characterize the neurophysiological (TMS) and brain signaling (EEG) profile of patients and specific muscles that respond to the combination of neuromodulation and robotic motor training.

DETAILED DESCRIPTION:
Current training interventions for rehabilitating patients with SCI are designed to provide the greatest possible restoration of function in the shortest possible time. One of the major deficits in our current approach to applying therapy is that we have little ability to predict which patients are most likely to respond to therapy or which muscle groups are most amenable to improvement. Transcranial magnetic stimulation (TMS) is a noninvasive method to excite or inhibit neurons in the brain or the spinal cord. Numerous studies have been using this technique to map connections from the motor cortex via the spinal cord to peripheral muscles; and as a therapeutic tool to promote useful plasticity.

The significance of the present study lies in the potential of intensive upper limb motor training with a novel robotic device, in conjunction with transcranial direct current stimulation (tDCS) over the contralateral motor cortex, may enhance neural recovery and upper limb function in patients with tetraplegia.

The robotic training devices represent the most sophisticated interactive rehabilitation systems available on the current market; they are additionally appealing for their ability to quantify various aspects of movement, and they appear to be particularly powerful way to promote functional recovery. Furthermore, robotic devices can be used in collection of quantitative data from the patients, which can be interpreted to analyze their rate of progress. Rehabilitation robots are capable of providing important components of motor skill learning and muscle training: individually prescribed intensity, repetition, and performance feedback. Furthermore, they are a novel and reliable method of assessing voluntary motor control. Our center has extensive experience in the use of rehabilitation robotics in the assessment and training of voluntary motor control in SCI patients, as well as other neurological disorders. From the investigator's previous experience using robotic therapy in SCI patients they can predict that some patients (approximately 10%) will show direct benefits from the interactive robot training.

The use of neuromodulatory techniques (TMS, tDCS) has been used for the last 2 decades in neurorehabilitation with the aim of enhance motor recovery when paired with activity dependent plasticity (training). In this proposal the investigator's will be using a new tDCS device, StarStim® - a wireless multichannel device that allows EEG recording as well as real or sham tDCS stimulation.

The purpose of this study is: To explore the neurophysiological and electroencephalography (EEG) changes that one single session of tDCS and robotics has in the SCI population (Study 1); and to investigate upper limb motor recovery in chronic tetraplegia SCI patients, comparing two rehabilitation strategies: real or sham tDCS combined with upper-limb robotic therapy (Study 2), as well as to characterize the neurophysiological (TMS) and brain signaling (EEG) profile of patients and specific muscles that respond to the combination of neuromodulation and robotic motor training.

Study 1, Objective: To evaluate changes in cortical neurophysiological and biological brain signaling after a single session of tDCS. The TMS responses of the upper limb muscles with lack of voluntary motor control will be assessed prior and after 20 min of tDCS intervention. Additionally, the investigators will record EEG activity before, during and after the intervention.

Study 2, Objective: To explore the accumulative effects of 2 weeks of tDCS + Robotic training in cortical excitability and brain signaling. In addition, the investigators will investigate whether the intensive robotic training in conjunction with tDCS over the contralateral motor cortex area will enhance neural recovery and upper limb function in patients with tetraplegia.

The investigators will compare two different brain stimulation protocols to assess the enhancement of the motor performance of those muscles that lack motor control, comparing the effects of 2-weeks intensive hand-robotic training with real or sham tDCS.

The investigators hypothesize that the patients who undergo real tDCS in conjunction with prolonged intense robotic training will achieve greater improvements in motor function and sensation compared to their counterparts who are in the sham control group.

ELIGIBILITY:
Inclusion Criteria:

* Level of injury C5 to T1
* Chronic SCI > 6 months
* Tetraplegic with some degree of motor dysfunction in the upper limb
* Motor Incomplete/Complete
* Medically stable

Exclusion Criteria:

* < 6 month after injury
* History of head trauma and/or cognitive deficit
* History of stroke, seizures or other intracranial disease
* Medically unstable
* Concomitant neurological disorder
* Pre-existing medical conditions interfering with unrestricted movement of the hand/arm (e.g. osteoarthritis, injury to the joints)
* Inability to provide informed consent
* Contraindications for non-invasive brain stimulation (NIBS) techniques (TMS & tDCS)- see below.

Non-Invasive Brain Stimulation Contraindications

* Surgically implanted foreign bodies such as a pacemaker, implanted medication pump, metal plate in the skull
* Metal inside the skull (other than dental appliances or fillings) that may pose a physical hazard during magnetic stimulation.
* No skin condition
* Any significant medical or psychiatric illness
* History of epilepsy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2018-06-27 (Actual)

PRIMARY OUTCOMES:
Motor Threshold | Change in motor threshold from baseline to immediately post-intervention. This measure will also be repeated at a 1 month follow up evaluation.
  The necessary stimulator output to evoke a response in the target muscle
Action Research Arm Test | Baseline, immediately after intervention.
  Assessment of upper extremity motor improvements
Amplitude of Response | Change in amplitude from baseline to immediately post-intervention. This measure will also be repeated at a 1 month follow up evaluation.
  The size of the wave form (response) generated during motor threshold determination.

SECONDARY OUTCOMES:
Transcranial magnetic stimulation mapping | Baseline, immediately after intervention, and 1 month follow up
  Method of determining a specific muscle's spatial representation in the cortex.
Electroencephalography (EEG) Recording | Baseline, immediately after intervention, and 1 month follow up
  Assessment of electrical activity in the brain over a period of time, as determined non-invasively through electrodes placed on the head.
Muscle Strength Evaluation | Baseline, immediately after intervention, and 1 month follow up
  Maximum voluntary contraction of the studied upper extremity muscle
Upper Extremity Motor Score (UEMS) | Baseline, immediately after intervention
  Measure of upper extremity strength
Spinal Cord Independence Measure (SCIM III) | Baseline, immediately after intervention
  Measure of functional independence in activities of daily living
Visual Analogue Scale | Baseline, immediately after intervention
  Used as a self-report of pain
Quadriplegia Index of Function (QIF) | Baseline, immediately after intervention
  Quality of life scale
Jebsen-Taylor Hand Function Test | Baseline, immediately after intervention
  Assessment of fine motor skills
Motor Evoked Potential Facilitation | Baseline, immediately after intervention, and 1 month follow up
  Method of assessing a nerves response to an external stimuli (transcranial magnetic stimulation)

CONTACTS AND LOCATIONS:
Overall Officials: Mar Cortes, MD, Principal Investigator — Mt Sinai School of Medicine
Locations (1):
- Burke Medical Research Institute, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers at this time.

REFERENCES:
- [Background] Barbeau H, Nadeau S, Garneau C. Physical determinants, emerging concepts, and training approaches in gait of individuals with spinal cord injury. J Neurotrauma. 2006 Mar-Apr;23(3-4):571-85. doi: 10.1089/neu.2006.23.571. PMID 16629638
- [Background] Behrman AL, Harkema SJ. Physical rehabilitation as an agent for recovery after spinal cord injury. Phys Med Rehabil Clin N Am. 2007 May;18(2):183-202, v. doi: 10.1016/j.pmr.2007.02.002. PMID 17543768
- [Background] Krebs HI, Volpe B, Hogan N. A working model of stroke recovery from rehabilitation robotics practitioners. J Neuroeng Rehabil. 2009 Feb 25;6:6. doi: 10.1186/1743-0003-6-6. PMID 19243615
- [Background] Spooren AI, Janssen-Potten YJ, Kerckhofs E, Seelen HA. Outcome of motor training programmes on arm and hand functioning in patients with cervical spinal cord injury according to different levels of the ICF: a systematic review. J Rehabil Med. 2009 Jun;41(7):497-505. doi: 10.2340/16501977-0387. PMID 19543659
- [Background] Wirth B, Van Hedel HJ, Curt A. Changes in corticospinal function and ankle motor control during recovery from incomplete spinal cord injury. J Neurotrauma. 2008 May;25(5):467-78. doi: 10.1089/neu.2007.0472. PMID 18419251
- [Background] Yozbatiran N, Berliner J, O'Malley MK, Pehlivan AU, Kadivar Z, Boake C, Francisco GE. Robotic training and clinical assessment of upper extremity movements after spinal cord injury: a single case report. J Rehabil Med. 2012 Feb;44(2):186-8. doi: 10.2340/16501977-0924. PMID 22334347